CLINICAL TRIAL: NCT01954602
Title: A Multicenter Randomized Trial Comparing the Use of Touch and no Touch Guide-wire Techniques for Deep Biliary Cannulation: the TNT Study
Brief Title: Use of Touch and no Touch Guide-wire Techniques for Deep Biliary Cannulation: the TNT Study
Acronym: TNT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Usl di Bologna (Other Government)
Collaborators: Catania Hospital Gastroenterology (Unknown); Niguarda Hospital (Other)
Responsible Party: Principal Investigator, CARLO DESCOVICH, Medical Doctor, Azienda Usl di Bologna
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CE 13028 TNT study
Record Dates: First submitted 2013-08-05; First posted 2013-10-07 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Biliary Tract Diseases
Keywords: Biliary cannulation; Endoscopic retrograde cholangiopancreatography; Touch guide-wire techniques; No touch guide-wire techniques
MeSH Terms: conditions — Biliary Tract Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Touch group (Active Comparator): Sphincterotome assisted guide-wire cannulation
  Interventions: Procedure: Sphincterotome assisted guide-wire cannulation
- No touch group (Experimental): Guide-wire cannulation
  Interventions: Procedure: Guide-wire cannulation

INTERVENTIONS:
Procedure: Guide-wire cannulation — Direct guide-wire hovering a few millimeters through the catheter or sphincterotome
  Arms: No touch group
Procedure: Sphincterotome assisted guide-wire cannulation — Sphincterotome is inserted initially a few millimeters through the papillary orifice
  Arms: Touch group

SUMMARY:
The specific goal of this study is to compare the deep biliary cannulation rate and complication rates associated with use of touch and no touch guide-wire biliary cannulation techniques.

DETAILED DESCRIPTION:
The most common technique used to achieve primary deep biliary cannulation is the standard contrast-assisted method, in which a catheter or sphincterotome is introduced into the papilla in the direction of the bile duct and a contrast medium injected to confirm that the duct has been cannulated.

The biliary guidewire cannulation technique consists of the introduction of a guide-wire into the bile duct instead of contrast injection as the first maneuver.

The benefit of this technique, compared with classic contrast cannulation, has been demonstrated in several studies which show similar results and have been analyzed in a recent meta-analysis, including 5 studies and 1762 patients, and demonstrating that the use of the guide-wire technique significantly improved the primary cannulation rate from 74.9% to 85.3%. More importantly, significantly reduced the incidence of PEP from 8.6% to 1.6%.

There are several variations of this technique; the tip of the sphincterotome is inserted initially a few millimeters through the papillary orifice and then introduce the guide-wire to the target ("touch technique"). Another variation is direct cannulation with the guide-wire hovering a few millimeters through the catheter or sphincterotome ("no touch technique").

To date, there are no randomized controlled trials comparing the two above described way to access to biliary duct regarding efficacy and rate of complications.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Clinical symptoms, laboratory findings and radiological evidences of biliary disease
* Willing and able to comply with the study procedures and provide written informed consent to participate in the study

Exclusion Criteria:

* Age <18 yars
* Patients with previous sphincterotomy
* Patients with previous papillary endoscopic balloon dilation
* Presence of a previously placed plastic or metal biliary stent
* Presence of any esophageal or gastro/duodenal stent
* Pancreatic or ampullary cancer, proven by imaging and/or cytology and/or histology, are excluded as PEP is very uncommon in these subgroups and tumour-related anatomical variation may alter cannulation technique (consider substratify results for this subgroup, but exclude if duodenal stenosis precludes an attempt on the papilla)
* Patients with surgically altered anatomy (Bilroth II gastrectomy and Roux en Y anastomosis) are excluded as cannulation technique is fundamentally different from that in normal anatomy
* Presence of a diverticular papilla
* Presence of a duodenal stenosis
* Presence of a pancreas divisum
* Patients with contraindication to endoscopic procedures
* Hemodinynamic instability, any acute illness or exacerbation of chronic illness, acute infections.
* Platelet count less than 50,000/mm3 and INR no greater than 1.5 times upper limit of normal
* Inability or refusal to give informed consent.
* Refusal to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Cannulation success rate | No more than 5 minutes of biliary cannulation or 5 unintended pancreatic duct cannulation with the guidewire, with both techniques

SECONDARY OUTCOMES:
Incidences of PEP | from the intervention until two days

CONTACTS AND LOCATIONS:
Overall Officials: Elio Jovine, MD, Study Chair — AUSL Bologna
Locations (1):
- Azienda Unità Sanitaria Locale, Bologna, Bologna, Italy

REFERENCES:
- [Background] Rabenstein T, Schneider HT, Nicklas M, Ruppert T, Katalinic A, Hahn EG, Ell C. Impact of skill and experience of the endoscopist on the outcome of endoscopic sphincterotomy techniques. Gastrointest Endosc. 1999 Nov;50(5):628-36. doi: 10.1016/s0016-5107(99)80010-8. PMID 10536317
- [Background] Cotton PB, Lehman G, Vennes J, Geenen JE, Russell RC, Meyers WC, Liguory C, Nickl N. Endoscopic sphincterotomy complications and their management: an attempt at consensus. Gastrointest Endosc. 1991 May-Jun;37(3):383-93. doi: 10.1016/s0016-5107(91)70740-2. PMID 2070995
- [Background] Sherman S, Ruffolo TA, Hawes RH, Lehman GA. Complications of endoscopic sphincterotomy. A prospective series with emphasis on the increased risk associated with sphincter of Oddi dysfunction and nondilated bile ducts. Gastroenterology. 1991 Oct;101(4):1068-75. PMID 1889699
- [Background] Freeman ML, Nelson DB, Sherman S, Haber GB, Herman ME, Dorsher PJ, Moore JP, Fennerty MB, Ryan ME, Shaw MJ, Lande JD, Pheley AM. Complications of endoscopic biliary sphincterotomy. N Engl J Med. 1996 Sep 26;335(13):909-18. doi: 10.1056/NEJM199609263351301. PMID 8782497
- [Background] Loperfido S, Angelini G, Benedetti G, Chilovi F, Costan F, De Berardinis F, De Bernardin M, Ederle A, Fina P, Fratton A. Major early complications from diagnostic and therapeutic ERCP: a prospective multicenter study. Gastrointest Endosc. 1998 Jul;48(1):1-10. doi: 10.1016/s0016-5107(98)70121-x. PMID 9684657
- [Derived] Bassi M, Luigiano C, Ghersi S, Fabbri C, Gibiino G, Balzani L, Iabichino G, Tringali A, Manta R, Mutignani M, Cennamo V. A multicenter randomized trial comparing the use of touch versus no-touch guidewire technique for deep biliary cannulation: the TNT study. Gastrointest Endosc. 2018 Jan;87(1):196-201. doi: 10.1016/j.gie.2017.05.008. Epub 2017 May 18. PMID 28527615